CLINICAL TRIAL: NCT03886857
Title: Carry-over Effects of Transcutaneous Spinal Cord Stimulation for Spasticity Control on Inhibitory Circuits of the Spinal Cord: a Pilot Study
Brief Title: Segmental Mechanisms of Transcutaneous Spinal Cord Stimulation for Spasticity Control
Acronym: SCS_CorE_AT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Lackner (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor-Investigator, Peter Lackner, Chief Physician, Klinikum Floridsdorf
Organization: Klinikum Floridsdorf (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCS-CorE_AT
Record Dates: First submitted 2019-03-18; First posted 2019-03-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: transcutaneous spinal cord stimulation — noninvasive electrical stimulation of the human lumbar spinal cord

SUMMARY:
The aim of the pilot study is to gain first insights into the interaction of transcutaneous spinal cord stimulation with the altered activity of intraspinal circuits associated with spinal spasticity. The main goal is to evaluate the validity of the chosen measures and to generate a data base for statistical planning of a subsequent clinical study.

ELIGIBILITY:
Inclusion Criteria:

written informed consent prior to participation

for participants with intact CNS:

• no previous neurological or musculoskeletal disorders

for participants with spinal cord injury:

* Spinal cord injury due to trauma
* ≥ 12 months post-spinal cord injury
* complete or incomplete spinal cord injury classified as grade C or D on the American Spinal Injury Association Impairment Scale (AIS)
* neurological level of spinal cord injury: C3-T10
* preserved tendon and cutaneo-muscular reflexes in the lower limbs

Exclusion Criteria:

* other neuromuscular diseases, e.g., amyotrophic lateral sclerosis (ALS), Parkinson's disease, Guillain-Barré syndrome, muscular dystrophy
* active implants (e.g., cardiac pacemaker, drug pump)
* passive implants at vertebral level T10 or caudal (e.g., metal screws/plates for surgical stabilization of spinal fractures)
* active infections or diseases, pressure sores
* dermatological issues at the stimulation site
* malignant diseases
* heart insufficiency (NYHA III-IV)
* potential pregnancy (pregnancy test to be conducted in women of child bearing age before application of transcutaneous spinal cord stimulation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Postsynaptic inhibition | pre-intervention to 2 hours post-intervention
  reciprocal inhibition of the soleus H-reflex

SECONDARY OUTCOMES:
Presynaptic inhibition | pre-intervention to 2 hours post-intervention
  induced D1 inhibition and ongoing presynaptic inhibition of the soleus-H reflex
H_max/M_max | pre-intervention to 2 hours post-intervention
  Ratio of the maximum H reflex and the maximum M wave
Low-frequency depression | pre-intervention to 2 hours post-intervention
  rate-dependent depression of the soleus H-reflex
Evaluation of lower-limb spasticity | pre-intervention to 2 hours post-intervention
  surface-electromyography based assessments

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Hofstoetter, Prof., PhD, Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Medical University of Vienna, Vienna
  - Klinik Floridsdorf, Vienna

IPD SHARING:
Plan to Share IPD: No